CLINICAL TRIAL: NCT02282085
Title: A Randomized, Multi-site, Parallel-group, Rater-blind Study Comparing Response With Aripiprazole Once Monthly and Standard of Care Oral Antipsychotics in Non-adherent Outpatients With Schizophrenia Identified Using the Brief Adherence Rating Scale
Brief Title: Treatment Study Comparing Aripiprazole Once Monthly With Standard of Care Medication in Outpatients With Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Matt Byerly (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Matt Byerly, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COL.AOM.2013.004
Record Dates: First submitted 2014-09-30; First posted 2014-11-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia
Keywords: Medication Non-Adherence; Antipsychotic
MeSH Terms: conditions — Schizophrenia; Medication Adherence | interventions — Antipsychotic Agents; Risperidone; Lurasidone Hydrochloride; Quetiapine Fumarate; Olanzapine; ziprasidone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole Once-Monthly (Experimental): Switch to 400 mg aripiprazole once-monthly injection
  Interventions: Drug: Aripiprazole Once-Monthly
- Standard of Care (Active Comparator): Continue current SOC oral antipsychotic medication
  Interventions: Drug: Oral Antipsychotic (i.e. aripiprazole, risperidone, lurasidone, quetiapine, olanzapine, ziprasidone, etc)

INTERVENTIONS:
Drug: Aripiprazole Once-Monthly
  Arms: Aripiprazole Once-Monthly
Drug: Oral Antipsychotic (i.e. aripiprazole, risperidone, lurasidone, quetiapine, olanzapine, ziprasidone, etc) — Oral antipsychotic medication
  Arms: Standard of Care

SUMMARY:
This study compares aripiprazole once-monthly injection to standard of care oral antipsychotic medication in non-adherent outpatients with schizophrenia to see which treatment helps people take their medicine more regularly and have more positive outcomes.

It is hypothesized that non-adherent schizophrenia outpatients receiving aripiprazole once-monthly will be more likely to respond and have lower symptom severity over 3 months of treatment than those receiving standard of care oral antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* Are able to provide written informed consent. If the Institutional Review Board (IRB) requires consent by a legally acceptable representative in addition to the subject, all required consents must be obtained prior to the initiation of any protocol-required procedure.
* Are 18 to 60 years of age, inclusive, at the time of informed consent
* Has a current diagnosis of schizophrenia, as defined by DSM-V criteria and a history of the illness for at least 6 months prior to screening from a reliable source (e.g., health care provider, family member, or medical records).
* Have been prescribed a single oral antipsychotic medication for at least 3 months prior to screening.
* Are able to understand the nature of the study and follow protocol requirements, including the prescribed dosage regimens, tablet ingestion, intramuscular (IM) once monthly injection, and discontinuation of prohibited concomitant medications, read and understand the written word in order to complete subject-reported outcomes measures, and be reliably rated on assessment scales.
* Are male and female subjects who are surgically sterile (i.e., have undergone orchiectomy or hysterectomy, respectively; female subjects who have been postmenopausal for at least 12 consecutive months; or male and female subjects who agree to remain abstinent or to practice double barrier forms of birth control from study screening through 30 days (for females) and 90 days (for males) from the last dose of study drug for SOC oral antipsychotics and 150 days for females and 180 days for males for aripiprazole once monthly. If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control implant, birth control once monthly injections, condom, or sponge with spermicide.

Exclusion Criteria:

* Has a current DSM-V diagnosis other than schizophrenia, including schizophreniform disorder, schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also excluded are subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Has had a psychiatric hospitalization within the 30 days prior to screening.
* Has received a depot antipsychotic within the 6 months prior to screening.
* Is considered resistant or refractory to antipsychotic treatment by history (failed two prior antipsychotic medication studies) or response only to clozapine.
* Is taking two or more antipsychotics.
* Has a significant risk of violent behavior or a significant risk of committing suicide based on history or investigator's discretion.
* Has a history of seizures or any other medical condition that would expose the subject to undue risk or interfere with study assessments.
* Is involuntarily incarcerated or has been incarcerated in the past 6 months for any reason.
* Has undergone electroconvulsive therapy in the 2 years prior to enrollment in the study.
* Has used an investigational agent or has participated in a clinical study with aripiprazole once monthly or any other antipsychotic once monthly preparation within 30 days of screening.
* Has any medical condition that might preclude safe completion of the study (e.g., agranulocytosis, severe and unstable heart disease, AIDS, end-stage renal disease).
* Is taking a CYP3A4 inducer (e.g., carbamazepine).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: PANSS (Positive and Negative Syndrome Scale) total score improvement - response | from date of randomization up to 3 months
  PANSS total score - operationalized as a binary response, defined as at least a 20% improvement in PANSS totals core, from the three monthly visits.

SECONDARY OUTCOMES:
Efficacy: PANSS total score overall - symptom severity | from date of randomization up to 3 months
  PANSS total score - continuous, from the three monthly visits
Quality of Life | from date of randomization up to 3 months
  Schizophrenia Quality of Life Scale (SQLS)
Cognition | from date of randomizatino up to 3 months
  Brief Assessment of Cognition in Schizophrenia (BACS)
Substance Use | from date of randomization up to 3 months
  Alcohol Use Scale (AUS) and Drug Use Scale (DUS)
Safety assessed by Treatment-emergent adverse events (TEAEs), physical examination including vital signs, clinical laboratory testing including prolactin and lipid profiles, and the Columbia Suicide Severity Rating Scale (C-SSRS) | from date of randomization up to 3 months
  Treatment-emergent adverse events (TEAEs), physical examination including vital signs, clinical laboratory testing including prolactin and lipid profiles, and the Columbia Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Byerly, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States